CLINICAL TRIAL: NCT02819219
Title: Effects of ElevATP on Body Composition and Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MusclePharm Sports Science Institute (Industry)
Collaborators: VDF FutureCeuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: VDFMPSSI01
Record Dates: First submitted 2016-06-22; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Dietary Supplements; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive a flavored water placebo supplement. Part of the supplemental intervention. This, and all groups, simultaneously took part in the exercise intervention.
  Interventions: Dietary Supplement: Supplemental; Other: Exercise Intervention
- ElevATP (Experimental): Participants will receive the flavored water placebo with an additional 150mg of ElevATP (blend of ancient peat and apple extracts). Part of the supplemental intervention.This, and all groups, simultaneously took part in the exercise intervention.
  Interventions: Dietary Supplement: Supplemental; Other: Exercise Intervention
- ElevATP w/Caffeine (Experimental): Participants will receive the flavored water placebo with an additional 150mg of ElevATP (blend of ancient peat and apple extracts), a 180 mg blend of caffeine (caffeine anhydrous, pterostilbene-bound caffeine), and 38mg B vitamins. Part of the supplemental intervention.This, and all groups, simultaneously took part in the exercise intervention.
  Interventions: Dietary Supplement: Supplemental; Other: Exercise Intervention

INTERVENTIONS:
Dietary Supplement: Supplemental — participants were provided with either placebo, placebo + ElevATP, or placebo + ElevATP + Caffeine + Vitamins.
  Other Names: ElevATP, PurEnergy
Other: Exercise Intervention — Concurrent with the supplemental intervention, all subjects participated in a resistance exercise intervention.

SUMMARY:
This study will examine the effects of supplemental ElevATP with or without a blend of extended-release caffeine and B vitamins for changes in body composition, athletic performance, and hematology over a 12 week intervention period.

DETAILED DESCRIPTION:
In a double-blind, placebo, diet, and training controlled design, 57 subjects will participate in an eight week, resistance and high intensity interval training study to assess the ergogenic potential of elevATP with and without caffeine plus vitamins in comparison to a visually identical, equal volume placebo within a periodized training program (described below). Prior to testing or training, subjects will report to the laboratory for screening and familiarization with testing protocols. The following week, subjects will complete baseline testing for all measurements including a 3 day food log. During the next eight weeks, subjects will participate in a periodized resistance training program which alters the repetition and loading schemes daily and weekly. During the entirety of the training protocol, subjects will supplement daily with either 1 serving of elevATP, 1 serving of Dropz (elevATP + caffeine), or 1 serving of an equal volume, visually identical placebo. Measurements will be repeated at the end of weeks 4 and 8, 10, and 12.

Variables collected:

* Dual Emissions X-Ray Absorptiometry (DEXA) determined (weeks 0, 4, 8, 10, 12):

  * Body fat
  * Lean body mass
  * Body fat percentage
* Bioelectric Impedance Analysis and Spectroscopy (BIA/BIS) determined (weeks 0, 4, 8, 10, 12):

  * Body fat
  * Lean body mass
  * Body fat percentage
* Ultrasonography determined cross-sectional area (weeks 0, 4, 8 , 10, 12)
* 1-repetition maximum (1RM) strength of the squat (weeks 0, 4, 8 , 10, 12)
* 1RM strength of the bench press (weeks 0, 4, 8 , 10, 12)
* 1RM strength of the deadlift (weeks 0, 4, 8 , 10, 12)
* Vertical jump height and power (weeks 0, 4, 8 , 10, 12)
* Bench press power (weeks 0, 4, 8 , 10, 12)
* Anaerobic peak and average power output (weeks 0, 4, 8 , 10, 12)
* Blood count, metabolic, and lipid safety panels (weeks 0, 8, and 12)
* Anthropometrics (weeks 0, 4, 8 , 10, 12)
* Vital Signs (weeks 0, 4, 8 , 10, 12)
* Myokines and biomarkers of regeneration panels (weeks 0, 4, 8, and 12): Analysis to be performed by VDF FutureCeuticals, Inc. MusclePharm to ship frozen serum samples (1-2ml) from all subjects to VDF FutureCeuticals, care of Zbigniew Pietrzkowski, 16259 Laguna Canyon Rd, Irvine, CA 92618

Resistance training protocol

Will consist of a daily undulating periodization design with high volume, high velocity, and high intensity workouts. Exercises performed will be the back squat, bench press, deadlift, leg press, bent row, shoulder press, pulldown, dips, bicep curl, tricep extension, single-arm row, hammer strength chest press, lateral raise, incline bench press, power squat, leg extension, and leg curl. Exercises will be performed for 1-15 repetitions, 3-5 sets, and with 0.5-5 minutes rest between sets.

Diet Each subject will receive a personalized diet to suit their individual needs. Total calories will be calculated based on the Mifflin St. Jeor equation. One half of total calories will be derived from carbohydrates, while fats and proteins will equally compose the remaining one half of total calories.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years
* Healthy as assessed by Pre-exercise Testing Health Status and General Information Questionnaire
* Strength trained for a minimum of 3 years as assessed by pre-exercise testing questionnaire
* Minimum strength requirements of 1x bodyweight bench press and 1.5x bodyweight squat and deadlift.
* Subject has provided written and dated informed consent to participate in the study

Exclusion Criteria:

* Having a history of medical events that may significantly affect the study outcome, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders
* Use of medicine that may significantly affect the study outcome
* Use of any ergogenic aids for one month prior to the onset of the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Fat (in kilograms) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by dual emissions x-ray absorptiometry (DEXA), bioelectric impedance analysis (BIA), and bioelectric impedance spectroscopy (BIS)
Change in Muscle Mass (in kilograms) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by dual emissions x-ray absorptiometry (DEXA), bioelectric impedance analysis (BIA), and bioelectric impedance spectroscopy (BIS)
Change in Body Fat percent (%) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by dual emissions x-ray absorptiometry (DEXA), bioelectric impedance analysis (BIA), and bioelectric impedance spectroscopy (BIS)
Change in Cross-sectional area of the rectus femoris (cm squared) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by ultrasound at 75% femur length.
Change in Maximal strength (in kilograms) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by 1-repetition maximum in the squat, bench press, and deadlift exercises.
Change in Power output (in watts) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by linear force transducer and cycle ergometer
Change in vertical jump height (in centimeters) | measure at 0, 4, 8, 10, and 12 weeks of the intervention
  Measured by vertec.

SECONDARY OUTCOMES:
Change in white blood cells (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in red blood cells (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in platelets (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in neutrophils (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in eosinophils (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in basophils (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in monocytes (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in lymphocytes. (number of cells per unit of blood volume) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, Laboratory Corporation of America (LabCorp)
Change in hemoglobin (grams per deciliter) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in mean corpuscular hemoglobin concentration (grams per deciliter) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in hematocrit (%) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in red blood cell distribution width (%) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in mean corpuscular volume (fL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in mean corpuscular hemoglobin (pg) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in serum glucose (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in blood urea nitrogen (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in creatinine (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in calcium (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in serum glucose, blood urea nitrogen, creatinine, calcium, total protein, albumin, globulin, bilirubin, total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein, and very low density lipoprotein (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in total protein (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in albumin (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in globulin (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in bilirubin (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in total cholesterol (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in triglycerides (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in high-density lipoprotein (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in low-density lipoprotein (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in very low density lipoprotein (mg/dL) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in estimated glomerular filtration rate (mL/min/1.73) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in serum sodium (mmol/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in serum potassium (mmol/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in serum chloride (mmol/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in serum carbon dioxide (mmol/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in aspartate aminotransferase (IU/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in alanine aminotransferase (IU/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in alkaline phosphatase (IU/L) | measure at 0, 8, and 12 weeks of the intervention
  measured by third party, LabCorp
Change in Irisin (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in Interleukin-6 (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in interleukin-15 (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in fibroblast growth factor-21 (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in myonectin (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in cortisol (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in c-reactive protein (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay
Change in growth differentiation factor-11 (pg/mL) | measure at 0, 4, 8, and 12 weeks of the intervention
  measured by enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: jordan m joy, ms, Principal Investigator — MusclePharm Sports Science Institute

IPD SHARING:
Plan to Share IPD: Undecided
The decision is not for the researchers to make and must consult with the funding agencies

REFERENCES:
- [Derived] Joy JM, Vogel RM, Moon JR, Falcone PH, Mosman MM, Pietrzkowski Z, Reyes T, Kim MP. Ancient peat and apple extracts supplementation may improve strength and power adaptations in resistance trained men. BMC Complement Altern Med. 2016 Jul 18;16:224. doi: 10.1186/s12906-016-1222-x. PMID 27430755